CLINICAL TRIAL: NCT03274453
Title: A Prospective, Randomized, Double Blinded Comparison of Ketamine Infusion Versus Placebo in Opioid Tolerant and Opioid Naive Patients After Spinal Fusion
Brief Title: A Comparison of Ketamine Infusion Versus Placebo in Opioid Tolerant and Opioid Naive Patients After Spinal Fusion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-02202
Record Dates: First submitted 2017-09-05; First posted 2017-09-07 (Actual); Results first posted 2018-06-14 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-05

CONDITIONS: Spinal Fusion
MeSH Terms: interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Ketamine Naive (Active Comparator): After an initial bolus of 0.2 mg/kg, the dose will be fixed at 0.12 mg/kg/hr of ketamine.
  Infusion will be maintained for 24 hours.
  Interventions: Drug: Ketamine
- Naive Placebo (Placebo Comparator): Saline will be administered at the same rate as the ketamine infusion. Infusion will be maintained for 24 hours.
  Interventions: Drug: Saline
- Tolerant Placebo (Placebo Comparator): Saline will be administered at the same rate as the ketamine infusion. Infusion will be maintained for 24 hours.
  Interventions: Drug: Saline
- Tolerant Ketamine (Experimental): After an initial bolus of 0.2 mg/kg, the dose will be fixed at 0.12 mg/kg/hr of ketamine.
  Infusion will be maintained for 24 hours.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — 0.12 mg/kg/hr of ketamine post surgery
  Arms: Ketamine Naive; Tolerant Ketamine
Drug: Saline — Saline will be administered at the same rate as the ketamine infusion.
  Arms: Naive Placebo; Tolerant Placebo

SUMMARY:
The aim of the proposed study is to examine the effectiveness of low dose postoperative ketamine infusion as an analgesic adjuvant to morphine pca in opioid tolerant and opioid naïve patients after major spine surgery. Primary endpoints of the study are to determine the effectiveness of postoperative ketamine infusion in for the reduction of postoperative pain and opioid requirements.

DETAILED DESCRIPTION:
Subjects aged 16 to 75, ASA I to III, scheduled for an elective lumbar fusion surgery of at least two levels under general anaesthesia, were prospectively studied. We defined opioid-tolerant as the daily use of opioid pain medication (oxycodone, morphine, hydromorphone, fentanyl, methadone, or tramadol) during the two weeks before surgery. Patients who did not fulfil that criterion were deemed to be opioid-naïve. Exclusion criteria were poorly controlled hypertension, severe cardiac or pulmonary disease, elevated intraocular pressure, severe hepatic or renal dysfunction, pregnancy, a history of psychiatric disorder, inability to speak English, inability to understand the numerical pain scale or to operate the patient-controlled analgesia pump, and known allergy to ketamine or hydromorphone.

Patients were allocated to the opioid-naïve or opioid-tolerant arm as defined above, and subsequently randomized into two groups, for a total of 4 groups: the opioid-naïve ketamine, the opioid-naïve placebo, the opioid-tolerant ketamine, and the opioid-tolerant placebo. Patients in each group were randomized to receive either a ketamine infusion (ketamine bolus 0.2 mg/kg over 30 minutes, started on arrival in post-anesthesia care unit (PACU), followed by a fixed-rate infusion of 0.12 mg/kg/h for 24 hours), or placebo (identical volume/rate of normal saline). Randomization within each group was performed by the study coordinator using a computer-generated random number list in a 1:1 ratio. Study medication and placebo were produced according to the randomization list in identical and consecutively numbered 250 mL bags. The pharmacist was not involved in patient care. Information about treatment was concealed but available for unblinding in case of acute complications. During the entire study period investigators performing the postoperative assessments, medical staff (nurse, anesthesiologist, and surgeon), and subjects were blinded to group allocation.

In all patients, general anesthesia was induced with propofol based on patient weight. Rocuronium 0.6 - 1.2 mg/kg was used to facilitate endotracheal intubation. Anesthesia was maintained with propofol (variable rate to maintain bispectral index (BIS) at a level acceptable for surgical anesthesia), desflurane <1.5% mixed of air and oxygen, fentanyl, sufentanil, hydromorphone and morphine at the discretion of the anesthetic staff. Blood pressure was maintained within 20% of baseline, and hypotension was treated at the discretion of the anesthetic staff with isotonic sodium chloride solution, hetastarch, ephedrine and phenylephrine intravenously.

Most patients received 1000 mg of IV acetaminophen at the end of surgery (see Table 2). NSAIDs were not used in the immediate perioperative period because of the surgeons' concern that they might impede bone healing and proper fusion.

For all patients, postoperative pain treatment during the first 24 hours consisted of standard care of IV patient controlled analgesia (PCA) with hydromorphone (0.2 mg/dose, lockout 6 min, maximum 2 mg/h), started on arrival in PACU. Preoperatively, the patients were educated by the nursing staff in the use of the PCA pump and the numerical pain scale. Rescue medication of IV hydromorphone 0.2 to 0.3 mg as needed was administered by a nurse with the goal to reduce the numerical pain score (NPS; 0 = no pain, 10 = worst imaginable pain) below 4. Opioid pain medication was restricted to hydromorphone in order to allow for valid comparison between the groups. After 24 hours, the PCA was discontinued and all patients were treated according to the surgical department's standard regimen. Diazepam 2 mg IV was administered for severe muscle spasms as needed.

Moderate to severe nausea or vomiting was treated with IV ondansetron 4 mg. If ondansetron was ineffective, IV metoclopramide 10 mg was administered.

All postoperative assessments were performed by the study investigators or trained nurses blinded to group allocation. Cumulative IV hydromorphone consumption was calculated from 0 to 24 hours postoperatively. NPS were recorded at arrival to PACU, then every 30 min during the first 2 hours, and then every 2 hours on the floor during the first 24 hours after surgery while patients were awake.

The primary outcome was cumulative hydromorphone consumption during the first 24h after surgery. Secondary outcome was NPS in the same time period. We also recorded central nervous system adverse events during the same period.

ELIGIBILITY:
Inclusion Criteria:

* Adult and teenage (>/=16) male or female who will undergo surgery for multilevel (>4 level) spinal fusion from a posterior approach with general anesthesia, and who are fluent English speakers such that they can complete the pain score and satisfaction questionnaires whose scores are a critical outcome variable.
* If female, subject is non-lactating and is either:
* Not of childbearing potential
* Of childbearing potential but is not pregnant at time of baseline as determined by pre-surgical pregnancy testing.
* Subject is ASA physical status 1, 2, or 3.

Exclusion Criteria:

* anxiety
* psychiatric disorder
* Allergy or sensitivity to ketamine or dilaudid
* Deemed un-acceptable by study team
* Cognitively impaired (by history)
* Subject requires chronic antipsychotic medication
* Subject known to be in liver failure
* Subject for whom opioids or ketamine are contraindicated
* Patients with narrow angle glaucoma
* Patients with a history of psychosis

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2012-11-01 (Actual); Primary Completion 2014-11-01 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Boenigk, MD, Principal Investigator — Kirsten.Boenigk@nyumc.org
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Boenigk K, Echevarria GC, Nisimov E, von Bergen Granell AE, Cuff GE, Wang J, Atchabahian A. Low-dose ketamine infusion reduces postoperative hydromorphone requirements in opioid-tolerant patients following spinal fusion: A randomised controlled trial. Eur J Anaesthesiol. 2019 Jan;36(1):8-15. doi: 10.1097/EJA.0000000000000877. PMID 30113350

RESULTS

PARTICIPANT FLOW:
Groups:
- Naive Placebo; Tolerant Placebo: Saline will be administered at the same rate as the ketamine infusion.
- Naive Ketamine; Tolerant Ketamine: After an initial bolus of 0.2 mg/kg, the dose will be fixed at 0.12 mg/kg/hr of ketamine.
  Infusion will be maintained for 24 hours.
Period: Overall Study
Arm/Group | Naive Placebo | Naive Ketamine | Tolerant Placebo | Tolerant Ketamine
Started | 38 | 30 | 32 | 29
Completed | 34 | 24 | 28 | 25
Not Completed | 4 | 6 | 4 | 4
Not completed — Lost to Follow-up | 2 | 5 | 4 | 1
Not completed — Physician Decision | 2 | 0 | 0 | 3
Not completed — Surgery Cancelled | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naive Placebo | Naive Ketamine | Tolerant Placebo | Tolerant Ketamine | Total
Number analyzed (Participants) | 34 | 24 | 28 | 25 | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 34 | 24 | 28 | 25 | 111
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Male | 15 | 11 | 14 | 13 | 53
  Sex: Female | 19 | 13 | 14 | 12 | 58

OUTCOME MEASURES:

1. Primary Outcome: Hydromorphone Use/24 Hours postOP in mg/kg
Description: Hydromorphone use during the first postoperative 24 hours in mg/kg
Time Frame: 24 Hours
Measure: Mean (Inter-Quartile Range); unit: mg/kg
Arm/Group | Naive Placebo | Naive Ketamine | Tolerant Placebo | Tolerant Ketamine
Number analyzed (Participants) | 34 | 24 | 28 | 25
mg/kg | .13 [.06 to .18] | .09 [.05 to .15] | .27 [.2 to .37] | .19 [.16 to .24]

ADVERSE EVENTS:
Time Frame: 24 hours
Description: Patients were systematically asked about side effects such as headaches, confusion, anxiety, excessive sedation and blurry vision when seen at 24 hours postoperatively. The records were also searched for evidence of such side effects.
Arm/Group | Naive Placebo | Naive Ketamine | Tolerant Placebo | Tolerant Ketamine
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/24 | 0/28 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/24 | 0/28 | 0/25
Other Adverse Events (participants affected / at risk) | 0/34 | 0/24 | 0/28 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes